CLINICAL TRIAL: NCT04625296
Title: Behaviour and Experience of Communities Healthcare Professionals Facing the SARS CoV-2 Epidemic
Brief Title: Behaviour and Experience of Communities Healthcare Professionals Facing the SARS CoV-2 (COVID-19) Epidemic
Acronym: COVecu
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AP-HP 200512
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Healthcare Worker Facing COVID-19
Keywords: Healthcare worker ,; COVID-19; behaviour
MeSH Terms: conditions — COVID-19; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare professional: Communities Health professionals (doctors, nurses, physiotherapist) Working in the city, In metropolitan France, Having managed patients with COVID-19
  Interventions: Behavioral: Semi-directive interview; Behavioral: Questionnaire : Preparedness for Caregiving Scale

INTERVENTIONS:
Behavioral: Semi-directive interview — Semi-directive interview, lasting a maximum of 45 minutes
Behavioral: Questionnaire : Preparedness for Caregiving Scale — Preparedness for Caregiving Scale - 8 questions

SUMMARY:
The purpose of this study is to identify behaviours and experiences of communities healthcare professionals (doctors, nurses and physiotherapists) in the management of the SARS-CoV 2 epidemic by identifying the impact of the epidemic on their work, their personal life and the difficulties they had experienced.

DETAILED DESCRIPTION:
Given the overcrowding in hospital services, the management of the health crisis linked to the SARS-CoV-2 epidemic relies in particular on the Territorial Professional Health Communities, which include doctors, nurses and physiotherapists. The challenge of caring for patients in a health system described as suffering, raises questions about the experience of the epidemic at all levels of action. To our knowledge, there is no information to date on the experience of the health crisis of urban health professionals in terms of the impact on their professional and personal lives and the difficulties encountered.

Using a mixed, cross-sectional, observational and multicentric methodology, the aim of this study, lasting a total of 12 months, is to identify the impact on professional and personal life as well as the difficulties experienced by doctors, nurses and physiotherapists working in private practice in connection with a CPTS involved in the management of the health crisis.

Semi-directive interviews, lasting a maximum of 45 minutes, will be carried out with doctors, nurses and physiotherapists integrated into a CPTS and digitally recorded audio digitally and then transcribed literally and in full. They will be conducted by the researcher participating in the study. The transcribed interviews will be anonymised and kept in an office of the Clinical Research Unit Paris Centre in order to carry out the analysis as the interviews are carried out. Following the interview, the participant will be asked to answer the "Preparedness for Caregiving Scale" composed of 8 questions, each evaluated by a 4-level Likert scale. Over a planned inclusion period of 3 months, 75 health professionals (25 doctors, 25 nurses, 25 physiotherapists) will be included. The evaluation criteria of the study will be: i) The diversity of themes extracted during the analysis of the interviews, leading after analysis to a set of meta-themes describing all the experience stories ii) The score on 24 of the "Preparedness for Caregiving Scale".

This study will allow an enrichment of knowledge about the impact of the health crisis on professional and personal life and the difficulties encountered by urban health professionals (doctors, nurses and physiotherapists). But also the identification of the key needs of self-employed health professionals in the management of a health crisis, both in terms of health care skills and in terms of organisation and communication between the various players. Finally, this study will make it possible to identify the traumas experienced and/or felt by self-employed health professionals and the possible consequences of these traumas.

ELIGIBILITY:
Inclusion Criteria:

* Communities Health professionals (doctors, nurses, physiotherapist)
* Be integrate to a Territorial Professional Health Communities (TPHC)
* Having managed patients during the COVID-19 epidemic

Exclusion Criteria:

* Health professionals working in the hospital sector
* Health Students (medical, nursing, physiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of healthcare workers will be selected through Territorial Professional Health Communities (TPHC). These TPHC are organizations designed around a health project and formed on the initiative of city health professionals based on a territory defined by the professionals themselves.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Diversity of themes extracted about care situations management of the COVID-19 epidemic. | 1 Day
  The greatest possible diversity of themes extracted during the analysis of interviews. Identifying the impact of the epidemic of healthcare worker, their personal life and the difficulties they had experienced

SECONDARY OUTCOMES:
Preparedness for caregiving scale (PCS) | 1 Day
  8 questions, each evaluated by a 4-level Likert scale (min 0; max 32) higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Flora DEVOS, Nurse MSC PhD, Study Director — APHP
Locations (1):
- URC/CIC Paris Centre, Paris, France